CLINICAL TRIAL: NCT07271758
Title: PROmega Pilot Study of Clinic-based DHA Blood Screening in Early Pregnancy
Acronym: PROmega
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00140664
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Nutrient Deficiency
Keywords: DHA; Omega-3 fatty acids; Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DHA blood screening (Experimental): Measurement of DHA as percent of total fatty acids in red blood cells
  Interventions: Other: DHA blood screening

INTERVENTIONS:
Other: DHA blood screening — Measure of DHA as percent of total fatty acids in red blood cells

SUMMARY:
This pilot study will explore feasibility of routine implementation of the recommended blood-based screening of DHA status in early pregnancy in routine clinical care.

DETAILED DESCRIPTION:
This pilot study will be conducted within the Atrium Health Wake Forest Baptist general academic obstetric practice that serves patients in six clinic locations in the Winston-Salem area. The study will train clinical staff on the prenatal omega-3 evidence; work with Epic IT to add the DHA blood test to the early prenatal lab order set; provide screening results with interpretation to patients and clinicians via Epic; monitor uptake of screening and viewing of results; and review screening results and characteristics of screened patients. This pilot data will inform the design of a cluster randomized trial to compare DHA blood screening with US usual care on preterm birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients initiating prenatal care at participating clinics who are eligible for early pregnancy blood testing per American College of Obstetricians and Gynecologists (ACOG) standards

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Screening uptake percentage | First 20 weeks of pregnancy
  Percent of eligible patients who receive DHA screening

OTHER OUTCOMES:
Clinical staff training percentage | 60 days from activation
  Percent of eligible clinical staff completing training
Docosahexaenoic Acid (DHA) status | up to week 20 gestation
  Percent of screened patients with low DHA (<5% of total fatty acids)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sauder, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Sharing data is outside the scope of this pilot study.